CLINICAL TRIAL: NCT06419088
Title: Effect of Preoperative Individualized Education on Anxiety and Recovery in Patients Undergoing Minimally Invasive Lung Surgery
Brief Title: Effect of Preoperative Individualized Education on Anxiety and Recovery.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPIEAR
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Education
Keywords: Preoperative education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individualized education group (Other): received individualized educational interventions utilizing audiovisual materials
  Interventions: Other: Preoperative individualized education
- standard education group (No Intervention): only routine preoperative education

INTERVENTIONS:
Other: Preoperative individualized education — Based on the identified individual education needs, the researcher implemented audio-visual education to the intervention group in the ward.
  Arms: individualized education group

SUMMARY:
Researchers aim to investigate whether individualized preoperative education for patients is beneficial in reducing perioperative anxiety, promoting postoperative recovery, and enhancing postoperative quality of life. The educational content will cover aspects such as the surgery procedure, anesthesia, postoperative pain and anxiety management, recovery time, and any potential required treatments. All participants will be administered a questionnaire before the surgery to evaluate their specific concerns and fears. The intervention group will receive preoperative education through audio-visual materials followed by targeted preoperative counseling, while the control group will receive routine preoperative education.

DETAILED DESCRIPTION:
Patients who met the research criteria were consulted prior to surgery, during which the research objectives were explained, and written consent was obtained. Following baseline assessment, patients were randomly allocated to either the individualized education group or the routine education group. Sociodemographic information was collected through face-to-face interviews conducted in the ward. Additionally, levels of anxiety and adverse events (sleep, pain, nausea, vomiting) were measured using the Visual Analog Scale (VAS) and Hospital Anxiety and Depression Scale (HADS). Patient anxieties regarding different aspects were assessed using specific concerns and fears scales.

The intervention group received individualized educational interventions utilizing audiovisual materials. Based on identified personalized educational needs, researchers administered individualized preoperative education to the intervention group in the ward. Patients in the control group received only routine preoperative education from clinical nurses.

The second assessment was conducted before patients were transferred to the operating room. Anxiety levels and adverse events (preoperative sleep, pain, nausea, and vomiting) were assessed using HADS and VAS. Postoperatively, pain, nausea, vomiting, and coughing were evaluated three times daily for the first three days (every 8 hours) using the Visual Analog Scale (VAS), and sleep was assessed daily using the Athens Insomnia Scale (AIS). Chronic symptoms and quality of life were assessed at postoperative weeks 1, 2, 4, 12, 26, and 52. Chronic cough was evaluated using the Leicester Cough Questionnaire, and chronic pain was evaluated using the Brief Pain Inventory. The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) and HADS were used for continuous assessment of quality of life, anxiety, and depression status.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above;
2. Received single-port thoracoscopic surgery;
3. Volunteered to participate in the study and signed an informed consent form.

Exclusion Criteria:

1. Presence of a mental disorder
2. Preoperative pain
3. Pregnancy
4. Presence of other tumours requiring treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety status | Before and after education, 12 months after surgery
  Change in anxiety intensity scores
Postoperative pain | Baseline, postoperative days 1,2,3
  The Visual Analog Scale (VAS) was used to evaluate the intensity of pain, where 0 meant no pain, and 10 - the most severe pain.
Postoperative nausea and vomiting | Baseline, postoperative days 1,2,3
  The Visual Analog Scale (VAS) was used to evaluate the intensity of nausea and vomiting
Sleep disorders | Baseline, postoperative days 1,2,3
  Change in Athens Insomnia Scale

SECONDARY OUTCOMES:
Postoperative Complications | 12 months after surgery
  The incidence of common postoperative complications
Quality of life after surgery | Baseline, 12 months after surgery
  Change from baseline in quality of life scores on the European Organisation for Research and Treatment of Cancer 30 item Quality of Life Questionnaire at postoperative weeks 1, 2, 4, 12, 26, and 52.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chen, Prof, Study Chair — Key Laboratory of Cardio-Thoracic Surgery, Fujian Medical University, Fujian Province University, Fu
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No